CLINICAL TRIAL: NCT06102863
Title: Progesterone Therapeutic Regimen Plus Statins in Young Women With Early Endometrial Carcinoma and Atypical Endometrial Hyperplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beihang University (Other); Peking University (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Secretary of the Party Committee,Vice president, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20231022
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Atypical Endometrial Hyperplasia and Endometrial Carcinoma Stage I
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Patients with endometrial cancer who met the inclusion criteria were randomly divided into the control group and the experimental group in a 1:1 ratio according to the random numbers generated in advance (no preset position, no specific object).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or mirena +GnRHa 3.75mg subcutaneous injection monthly);
- experimental group (Experimental): Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with statins (oral atorvastatin calcium tablet 20mg/ day; Or rosuvastatin 5mg/ day; Or pivastatin 2mg/ day);
  Interventions: Drug: statins (oral atorvastatin calcium tablet 20mg/ day; Or rosuvastatin 5mg/ day; Or pivastatin 2mg/ day);

INTERVENTIONS:
Drug: statins (oral atorvastatin calcium tablet 20mg/ day; Or rosuvastatin 5mg/ day; Or pivastatin 2mg/ day); — Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with statins (oral atorvastatin calcium tablet 20mg/ day; Or rosuvastatin 5mg/ day; Or pivastatin 2mg/ day);
  Arms: experimental group

SUMMARY:
To explore the treatment efficacy of Progesterone Therapeutic Regimen Plus Statins in patients with atypical endometrial hyperplasia (AEH) and early endometrial carcinoma (EEC) for conservative treatment.

DETAILED DESCRIPTION:
After diagnosed of AEH or EEC by hysteroscopy, patients meet the study criteria will be enrolled. The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion tissue was detected by Raman scattering instrument. And Age, height, weight, waistline, blood pressure, basic history of infertility and family cancer will be collected. Blood tests, including fasting blood glucose (FBG), fasting insulin (FINS), blood lipids, sex hormone levels, anti-müllerian hormone (AMH) and renal/liver function tests will be performed before treatment to evacuate their basic conditions. Each subject will receive body fat testing by Inbody 770.

Patients with endometrial cancer who met the inclusion criteria were randomly divided into the control group and the experimental group in a 1:1 ratio according to the random numbers generated in advance. The administration regimen for the two groups was as follows:

1. Control group: progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa 3.75mg subcutaneous injection monthly);
2. Trial group: progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with statins (oral atorvastatin calcium tablet 20mg/ day; or rosuvastatin 5mg/ day; or pivastatin 2mg/ day);

The specific selection of progesterone regimen was based on whether the patients had oral progesterone contraindications and if BMI≥28kg/m2 was not suitable for oral progesterone, Mirena +GnRHa regimen was selected. The choice of statin drugs is based on the results of the drug sensitivity test of the patient's tumor tissue, and the most sensitive one of the three drugs is selected.

For patients remained SD after 9 months of treatment but refused hysterectomy, a multiple disciplinary discussion would be held for individual case, and alternative treatment would be given. Maintenance treatment will be recommended for patients with CR, and participants will be followed up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* The pathological types are consistent with:

  1. Atypical endometrial hyperplasia;
  2. Patients with highly differentiated endometrioid adenocarcinoma, stage IA, and pelvic and abdominal MRI before treatment excluded deep muscle infiltration, cervical involvement, and extrauterine metastasis;
  3. There is a strong need to preserve reproductive function; Age ≤45 years old;
  4. Progesterone resistant patients predicted by the progesterone sensitivity prediction model (NCT05647109) established by our team in the previous study of endometrial cancer were prospectively randomized; The predicted progesterone sensitive patients were prospectively observed;
  5. Informed consent and signed informed consent;
  6. have follow-up conditions and are willing to continue to follow the visitors in the hospital;
  7. Patients with normal/abnormal blood lipids who have not taken any lipid-lowering drugs;
  8. A. Newly treated patients: did not use any nursery therapy drugs (progesterone, GNRH-a); B. 1 course of treatment (12 weeks) the lesions persisted; C. Partial remission for 2 courses of treatment (24 weeks);

Exclusion Criteria:

* (1) Patients with severe internal diseases and severe impairment of liver and kidney function;

  (2) Disease progression, extrauterine metastasis (cervical invasion or distant metastasis such as pelvic cavity) during treatment;

  (3) People with therapeutic drug allergies and contraindications;

  (4) Patients with other types of endometrial cancer or other malignant tumors of the reproductive system; Patients with breast cancer or other hormone-dependent tumors that cannot use progesterone;

  (5) Patients with deep vein thrombosis, stroke and myocardial infarction during treatment;

  (6) Alcoholics (> 20g/ day);

  (7) Smokers (> 15 cigarettes/day)

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological cumulative complete response rate; | assessed up to 7 months
  From 6 to 7 months: From date of initial therapy until the date of CR.

SECONDARY OUTCOMES:
Pathological cumulative complete response rate; | assessed up to 4 months
  From 3 to 4 months; From date of initial therapy until the date of CR.
The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion tissue | assessed up to 7 months
  The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion
Overall complete response rate | up to 2 years
  Pathological response duration
Relapse rate | up to 15 months after the end of treatment.
  Relapse rate
Toxic Side Effect | up to 3 months after the end of treatment.
  Toxicity evaluation according to CTCAE 5.0 version.
Pregnancy rate | up to 15 months after the end of treatment.
  Number of pregnancies after complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, professor, Study Director — Peking University /Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No